CLINICAL TRIAL: NCT01858727
Title: The Effect of Preoperative Warming on Postoperative Hypothermia in TURP Surgery
Brief Title: The Effect of Preoperative Warming on Postoperative Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, Dr. fatma kavak akelma, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESM0606
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Preventing Hypothermia; Perioperative Hypothermia
Keywords: forced-air; hypothermia; TUR-P surgery; core temperatures; prewarming; general anaesthesia
MeSH Terms: conditions — Hypothermia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- forced air warming group (Active Comparator): 30 minutes before the preoperative will use forced air warming.
  Interventions: Other: forced air warming group; Other: control group
- control group (No Intervention): do not active heating group

INTERVENTIONS:
Other: forced air warming group — 30 minutes before the preoperative will use forced air warming
  Arms: forced air warming group
Other: control group — do not heating group
  Arms: forced air warming group

SUMMARY:
36 patients American society of anesthesiology (ASA) physical status I,II and III undergoing general anesthesia for elective transurethral resection of the prostate (TUR-P) surgery will be included in the study. Patients will be randomized into two groups; first group(control group) and second group (forced-air warming). Resistive heating will start when patients are transferred to the operating room table; forced-air warming will start before preoperative 30 minute.

DETAILED DESCRIPTION:
The primary aim of this study was to compare the effect of prewarming on perioperative hypothermia in elderly patients undergoing TURP under general anesthesia. In addition, we aimed to evaluate the effects of prewarming on hemodynamic variables, PACU output time, tremor, patient comfort and satisfaction. The investigators plan to enroll 36 patients in 2 groups. Body temperature will be measured at the core temperature, hemodynamic variables. Shivering will be graded by visual inspection. Thermal discomfort scale, patient satisfaction will be evaluated. The investigators hypothesize will decrease the forced air prewarming incidence of perioperative hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-85 years undergoing general anesthesia for TURP surgery
* ASA physical status I and III patients
* Body mass index between 15 and 36 kg/m2
* General anesthesia time is 30-90 minutes

Exclusion Criteria:

* without written consent,
* inadequate Turkish comprehension,
* known impaired thermoregulation or thyroid disorders,
* severe hypertension (systolic blood pressure [SBP]>180 mmHg or diastolic blood pressure [DBP] > 110 mmHg in the operating suite admission),
* an angiotensin-converting enzyme inhibitor/angiotensin II receptor antagonist on the day of surgery,
* secondary hypertension (e.g., renal artery stenosis, pheochromocytoma, Cushing's syndrome),
* vascular disease,
* poor cutaneous perfusion,
* serious skin lesions
* baseline temperature ≥37.5°C (degrees centigrade)

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Perioperative measurements of core temperature (centigrade ° C) | 2-3 hours
  After the operation patients will be admitted to the PACU. Here, body temperature will be assessed and the incidence of hypothermic patients (body temperature < 36°C)will be measured.

SECONDARY OUTCOMES:
Evaluation of hemodynamic variables (arterial blood pressure) | 2-3 hours
  systolic blood pressure (SBP) in mmHg, diastolic blood pressure (DBP) in mmHg, mean arterial pressure (MAP) in mmHg will be measured.
Evaluation of hemodynamic variables (heart rate) | 2-3 hours
  heart rate (HR) in beats per minute will be measured.
Number of patients with postoperative shivering | 2-3 hours
  After the operation patients will be admitted to the PACU. Here, postoperative shivering will be measured and graded by visual inspection.

OTHER OUTCOMES:
To assess patient satisfaction | 12 hours
  patient satisfaction scale (using a Likert scale type (range, 1 to 7) verbally administered questionnaire for patient satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: fakelma 905327079113, Principal Investigator — Diskapi Teaching and Research Hospital
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Altindag, Turkey (Türkiye)